CLINICAL TRIAL: NCT01582217
Title: TRIAGE: Patients Undergoing Percutaneous Coronary Interventions to Improve Clinical Outcomes Through Optimal Platelet Inhibition
Brief Title: Patients Undergoing Percutaneous Coronary Intervention (PCI) Through Optimal Platelet Inhibition
Acronym: TRIAGE
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Daiichi Sankyo (Industry); Accumetrics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 12-0028; FWA # 00005656 and 00005651
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Percutaneous Coronary Intervention; Dual Antiplatelet Therapy; Aspirin; Clopidogrel
Keywords: Bleeding; Risk Score; Outcomes; Prasugrel
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SA + 5mg prasugrel: Prasugrel 5 mg group: Patients with Intermediate or high bleeding risks and PRU ≥ 230 are Prescribed 5mg of prasugrel daily along with aspirin.
- ASA + 10 mg prasugrel: Prasugrel 10 mg group: Patients with Low bleeding risk and high ischemia risk and PRU ≥ 230 are prescribed 10 mg of prasugrel daily along with aspirin.
- ASA + 75 mg clopidogrel daily: Clopidogrel 75 mg group (control): PRU ≤ 230; high bleeding risk or high ischemic risk; patients with active malignancy, age >75; Wt< 60kg with previous CVA or TA are prescribed 75 mg of clopidogrel daily along with aspirin.

SUMMARY:
The purpose of this study is to assess the the 1-year rates of ischemic and bleeding complications in patients whose dual antiplatelet therapy regimen post-PCI has been determined with the use of a clinical algorithm that includes both clinical risks and platelet reactivity while on chronic clopidogrel therapy.

DETAILED DESCRIPTION:
Prospective multicenter registry. Patients already on chronic dual antiplatelet therapy with aspirin and clopidogrel will be assessed for (1) clinical risks factors for future bleeding and ischemic complications, and (2) on-treatment platelet reactivity as measured by the VerifyNow P2Y12 assay (Accumetrics, Inc., San Diego, CA, USA). These will be considered by utilization of a clinical algorithm to determine the dual antiplatelet regimen post-PCI (aspirin in combination with 1. clopidogrel, 2. prasugrel 5mg daily, or 3. prasugrel 10mg daily).

ELIGIBILITY:
Inclusion Criteria:

* The subject has provided informed written.
* The subject must be ≥ 18 years of age (or minimum age as required by local regulations) at the time of enrollment.
* Patient is established on chronic clopidogrel therapy when he/she returns for PCI, and the components of DAPT are determined by the clinical decision algorithm as local standard of care.
* The subject is willing and able to cooperate with the study procedures and required follow-ups.

Exclusion Criteria:

* Patients with cardiogenic shock will be excluded.
* The subject is participating in an investigational device or drug study. Subject must have completed the follow up phase of any previous study at least 30 days prior to enrolment in this study.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in any of the participating sites who are on chronic clopidogrel treatment and return for PCI will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
MACE | 12 months
  Major adverse cardiac events (all-cause death, myocardial infarction and stent thrombosis)

SECONDARY OUTCOMES:
Rates of major bleeding | 12 months
  The rates of major bleeding in patients treated with a thienopyridine based on the clinical algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: George Dangas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States